CLINICAL TRIAL: NCT02586220
Title: Iodine Nutrition During Pregnancy and Related Neonatal Physical Development
Status: Completed | Type: Observational
Sponsor: qingya tang (Other)
Responsible Party: Sponsor-Investigator, qingya tang, Chief Physician, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Other Study IDs: XHEC-C-2015-003-2
Record Dates: First submitted 2015-09-23; First posted 2015-10-26 (Estimated); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Pregnancy; Iodine Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — spot urine sample of pregnant women
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- normal pregnant women: 150 normal pregnant women (28-32 weeks' gestation)
- pregnant women with gestational: 100 pregnant women with gestational diabetes (28-32 weeks' gestation)

SUMMARY:
Recent studies have found, in both developed and developing countries, there is still a considerable number of pregnant women in iodine deficiency status.Our overall aim is to monitor iodine status of pregnant women in China, and to examine the correlation between maternal urine iodine concentration (UIC) and newborn physical development level.

DETAILED DESCRIPTION:
Background: Recent studies have found, in both developed and developing countries, there is still a considerable number of pregnant women in iodine deficiency status. Our overall aim is to monitor iodine status of pregnant women in China, and to examine the correlation between maternal urine iodine concentration (UIC) and newborn physical development level.

Design: prospective cohort study

Methods: During August - December 2015,250 participants(28-32 weeks' gestation) were selected to participate in the study.The investigators collect the spot urine samples(n=750) once every two weeks.

Setting: Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine.

Participants: 150 normal pregnant women and 100 pregnant women with gestational diabetes (28-32 weeks' gestation) and their newborns were selected to participate the study.

ELIGIBILITY:
Inclusion Criteria:

* 22-35 years,
* 28-32 weeks' gestation,

Exclusion Criteria:

* a known history of thyroid disease in the non-pregnant state and previous.

Ages: 22 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: 250 pregnant women recruited from antenatal outpatient clinics in Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medicine, China.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
urinary iodine (UI) concentrations | up to three months

SECONDARY OUTCOMES:
thyroid stimulating hormone level of newborns | up to three months
daily iodine intake of pregnant women | up to three months
  Daily iodine intake was estimated using the total diet study approach

CONTACTS AND LOCATIONS:
Overall Officials: Qingya Tang, MMed, Principal Investigator — Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Locations (2):
- China (2):
  - Xinhua Hospital Affiliated to Shanghai Jiaotong University School of Medcine, Shanghai, Shanghai Municipality
  - Xinhua Hospital, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Luo Y, Kawashima A, Ishido Y, Yoshihara A, Oda K, Hiroi N, Ito T, Ishii N, Suzuki K. Iodine excess as an environmental risk factor for autoimmune thyroid disease. Int J Mol Sci. 2014 Jul 21;15(7):12895-912. doi: 10.3390/ijms150712895. PMID 25050783
- [Background] Konig F, Andersson M, Hotz K, Aeberli I, Zimmermann MB. Ten repeat collections for urinary iodine from spot samples or 24-hour samples are needed to reliably estimate individual iodine status in women. J Nutr. 2011 Nov;141(11):2049-54. doi: 10.3945/jn.111.144071. Epub 2011 Sep 14. PMID 21918061
- [Background] Als C, Helbling A, Peter K, Haldimann M, Zimmerli B, Gerber H. Urinary iodine concentration follows a circadian rhythm: a study with 3023 spot urine samples in adults and children. J Clin Endocrinol Metab. 2000 Apr;85(4):1367-9. doi: 10.1210/jcem.85.4.6496. PMID 10770167
- [Background] Busnardo B, Nacamulli D, Zambonin L, Mian C, Piccolo M, Girelli ME. Restricted intraindividual urinary iodine concentration variability in nonfasting subjects. Eur J Clin Nutr. 2006 Mar;60(3):421-5. doi: 10.1038/sj.ejcn.1602334. PMID 16391581
- [Background] Knudsen N, Christiansen E, Brandt-Christensen M, Nygaard B, Perrild H. Age- and sex-adjusted iodine/creatinine ratio. A new standard in epidemiological surveys? Evaluation of three different estimates of iodine excretion based on casual urine samples and comparison to 24 h values. Eur J Clin Nutr. 2000 Apr;54(4):361-3. doi: 10.1038/sj.ejcn.1600935. PMID 10745289
- [Background] Zimmermann MB. Iodine deficiency. Endocr Rev. 2009 Jun;30(4):376-408. doi: 10.1210/er.2009-0011. Epub 2009 May 21. PMID 19460960
- [Background] Vejbjerg P, Knudsen N, Perrild H, Laurberg P, Carle A, Pedersen IB, Rasmussen LB, Ovesen L, Jorgensen T. Thyroglobulin as a marker of iodine nutrition status in the general population. Eur J Endocrinol. 2009 Sep;161(3):475-81. doi: 10.1530/EJE-09-0262. Epub 2009 Jun 25. PMID 19556382
- [Background] van den Briel T, West CE, Hautvast JG, Vulsma T, de Vijlder JJ, Ategbo EA. Serum thyroglobulin and urinary iodine concentration are the most appropriate indicators of iodine status and thyroid function under conditions of increasing iodine supply in schoolchildren in Benin. J Nutr. 2001 Oct;131(10):2701-6. doi: 10.1093/jn/131.10.2701. PMID 11584093
- [Background] Travers CA, Guttikonda K, Norton CA, Lewis PR, Mollart LJ, Wiley V, Wilcken B, Eastman CJ, Boyages SC. Iodine status in pregnant women and their newborns: are our babies at risk of iodine deficiency? Med J Aust. 2006 Jun 19;184(12):617-20. doi: 10.5694/j.1326-5377.2006.tb00417.x. PMID 16803441
- [Background] Leung AM, Braverman LE. Consequences of excess iodine. Nat Rev Endocrinol. 2014 Mar;10(3):136-42. doi: 10.1038/nrendo.2013.251. Epub 2013 Dec 17. PMID 24342882
- [Background] Katz PM, Leung AM, Braverman LE, Pearce EN, Tomlinson G, He X, Vertes J, Okun N, Walfish PG, Feig DS. Iodine nutrition during pregnancy in Toronto, Canada. Endocr Pract. 2013 Mar-Apr;19(2):206-11. doi: 10.4158/EP12193.OR. PMID 23186967
- [Background] WHO Secretariat; Andersson M, de Benoist B, Delange F, Zupan J. Prevention and control of iodine deficiency in pregnant and lactating women and in children less than 2-years-old: conclusions and recommendations of the Technical Consultation. Public Health Nutr. 2007 Dec;10(12A):1606-11. doi: 10.1017/S1368980007361004. No abstract available. PMID 18053287
- [Background] Caldwell KL, Makhmudov A, Ely E, Jones RL, Wang RY. Iodine status of the U.S. population, National Health and Nutrition Examination Survey, 2005-2006 and 2007-2008. Thyroid. 2011 Apr;21(4):419-27. doi: 10.1089/thy.2010.0077. PMID 21323596
- [Background] Perrine CG, Herrick K, Serdula MK, Sullivan KM. Some subgroups of reproductive age women in the United States may be at risk for iodine deficiency. J Nutr. 2010 Aug;140(8):1489-94. doi: 10.3945/jn.109.120147. Epub 2010 Jun 16. PMID 20554903
- [Background] Sullivan KM, Perrine CG, Pearce EN, Caldwell KL. Monitoring the iodine status of pregnant women in the United States. Thyroid. 2013 Apr;23(4):520-1. doi: 10.1089/thy.2012.0217. No abstract available. PMID 23157653
- [Background] Bath SC, Walter A, Taylor A, Wright J, Rayman MP. Iodine deficiency in pregnant women living in the South East of the UK: the influence of diet and nutritional supplements on iodine status. Br J Nutr. 2014 May;111(9):1622-31. doi: 10.1017/S0007114513004030. Epub 2014 Jan 7. PMID 24398008
- [Background] Zou S, Wu F, Guo C, Song J, Huang C, Zhu Z, Yu H, Guo Y, Lu X, Ruan Y. Iodine nutrition and the prevalence of thyroid disease after salt iodization: a cross-sectional survey in Shanghai, a coastal area in China. PLoS One. 2012;7(7):e40718. doi: 10.1371/journal.pone.0040718. Epub 2012 Jul 27. PMID 22911705
- [Background] Meng F, Zhao R, Liu P, Liu L, Liu S. Assessment of iodine status in children, adults, pregnant women and lactating women in iodine-replete areas of China. PLoS One. 2013 Nov 25;8(11):e81294. doi: 10.1371/journal.pone.0081294. eCollection 2013. PMID 24282581
- [Background] Alvarez-Pedrerol M, Guxens M, Mendez M, Canet Y, Martorell R, Espada M, Plana E, Rebagliato M, Sunyer J. Iodine levels and thyroid hormones in healthy pregnant women and birth weight of their offspring. Eur J Endocrinol. 2009 Mar;160(3):423-9. doi: 10.1530/EJE-08-0716. Epub 2008 Dec 29. PMID 19114540
- [Background] Rydbeck F, Rahman A, Grander M, Ekstrom EC, Vahter M, Kippler M. Maternal urinary iodine concentration up to 1.0 mg/L is positively associated with birth weight, length, and head circumference of male offspring. J Nutr. 2014 Sep;144(9):1438-44. doi: 10.3945/jn.114.193029. Epub 2014 Jul 16. PMID 25031330
- [Background] Olivares JL, Olivi GI, Verdasco C, Ortiz VA, Mayer MA, Cresto JC. Low iodine intake during pregnancy: relationship to placental development and head circumference in newborn. Endocrinol Nutr. 2012 May;59(5):326-30. doi: 10.1016/j.endonu.2011.12.005. Epub 2012 Feb 29. PMID 22381147
- [Background] Zhou SJ, Anderson AJ, Gibson RA, Makrides M. Effect of iodine supplementation in pregnancy on child development and other clinical outcomes: a systematic review of randomized controlled trials. Am J Clin Nutr. 2013 Nov;98(5):1241-54. doi: 10.3945/ajcn.113.065854. Epub 2013 Sep 11. PMID 24025628
- [Background] Rebagliato M, Murcia M, Alvarez-Pedrerol M, Espada M, Fernandez-Somoano A, Lertxundi N, Navarrete-Munoz EM, Forns J, Aranbarri A, Llop S, Julvez J, Tardon A, Ballester F. Iodine supplementation during pregnancy and infant neuropsychological development. INMA Mother and Child Cohort Study. Am J Epidemiol. 2013 May 1;177(9):944-53. doi: 10.1093/aje/kws333. Epub 2013 Apr 1. PMID 23548753
- [Background] Kevany J, Fierro-Benitez R, Pretell EA, Stanbury JB. Prophylaxis and treatment of endemic goiter with iodized oil in rural Ecuador and Peru. Am J Clin Nutr. 1969 Dec;22(12):1597-607. doi: 10.1093/ajcn/22.12.1597. PMID 4312017
- [Background] Pretell EA, Torres T, Zenteno V, Cornejo M. Prophylaxis of endemic goiter with iodized oil in rural Peru. Adv Exp Med Biol. 1972;30:246-65. No abstract available. PMID 4350937
- [Background] Pharoah PO, Connolly KJ. A controlled trial of iodinated oil for the prevention of endemic cretinism: a long-term follow-up. Int J Epidemiol. 1987 Mar;16(1):68-73. doi: 10.1093/ije/16.1.68. PMID 3032814
- [Background] Velasco I, Carreira M, Santiago P, Muela JA, Garcia-Fuentes E, Sanchez-Munoz B, Garriga MJ, Gonzalez-Fernandez MC, Rodriguez A, Caballero FF, Machado A, Gonzalez-Romero S, Anarte MT, Soriguer F. Effect of iodine prophylaxis during pregnancy on neurocognitive development of children during the first two years of life. J Clin Endocrinol Metab. 2009 Sep;94(9):3234-41. doi: 10.1210/jc.2008-2652. Epub 2009 Jun 30. PMID 19567536
- [Background] Berbel P, Mestre JL, Santamaria A, Palazon I, Franco A, Graells M, Gonzalez-Torga A, de Escobar GM. Delayed neurobehavioral development in children born to pregnant women with mild hypothyroxinemia during the first month of gestation: the importance of early iodine supplementation. Thyroid. 2009 May;19(5):511-9. doi: 10.1089/thy.2008.0341. PMID 19348584
- [Background] Hynes KL, Otahal P, Hay I, Burgess JR. Mild iodine deficiency during pregnancy is associated with reduced educational outcomes in the offspring: 9-year follow-up of the gestational iodine cohort. J Clin Endocrinol Metab. 2013 May;98(5):1954-62. doi: 10.1210/jc.2012-4249. Epub 2013 Apr 30. PMID 23633204
- [Background] Bath SC, Steer CD, Golding J, Emmett P, Rayman MP. Effect of inadequate iodine status in UK pregnant women on cognitive outcomes in their children: results from the Avon Longitudinal Study of Parents and Children (ALSPAC). Lancet. 2013 Jul 27;382(9889):331-7. doi: 10.1016/S0140-6736(13)60436-5. Epub 2013 May 22. PMID 23706508